CLINICAL TRIAL: NCT04481893
Title: Interest of the Virtual Reality Headset in the Management of Perioperative Stress in Patients Candidates for Total Thyroidectomy
Acronym: ThyroVir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A00182-37
Record Dates: First submitted 2020-07-07; First posted 2020-07-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer; Thyroidectomy
Keywords: virtual reality headset; stress; hypnose
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- using a virtual reality headset (Experimental)
  Interventions: Behavioral: Use of a virtual reality headset

INTERVENTIONS:
Behavioral: Use of a virtual reality headset — The intervention will consist of 2 sessions of 30 minutes each, based on the use of a virtual reality headset with the AQUA® application.
  * The 1st session will take place on the day of the surgical intervention, upon arrival in hospital, after reception in the room.
  * The 2nd session will take place the same day, post-operatively, once the awakening is satisfactory (within 3 to 6 hours after the intervention)

SUMMARY:
Study the interest of hypnosis techniques by virtual reality based on the use of a virtual reality headset with the AQUA® application on the reduction of pre-operative stress in patients candidates for total thyroidectomy

ELIGIBILITY:
Inclusion Criteria:

* Patient> 18 years old
* Man or woman
* Patient candidate for a total thyroidectomy, or a thyroid totalization
* Preoperative Euthyroidism
* Can justify outpatient care: score of the American Society of Anesthesiology (ASA) 1, 2 or 3 stable; accompanied for return at home; can be watched by a loved one the night after returning home; reachable by telephone; living within an hour of transportation from a hospital and having a good level of understanding.
* No history of parathyroid or recurrent pathology
* Signature of informed consent before any specific procedure related to the study
* Subject affiliated with a health security system

Exclusion Criteria:

* Patient with a submerged goiter (lower edge of the thyroid not seen on the preoperative cervical ultrasound)
* Patient with uncontrolled infectious pathology
* Pregnant or breastfeeding woman or lack of contraception during genital activity
* Patient with illnesses or conditions that hinder their ability to understand follow and / or comply with study procedures
* Patient with personality disorders and / or psychiatric pathology
* Patient deprived of liberty or placed under the authority of a guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Change of Anxiety state (STAI-Y scale) | Before surgery and up to 2 hours after surgery
  The proportion of patients whose pre-operative anxiety state (STAI-Y scale)is improved or stable between before and after the session with virtual reality headset. These two measurements will allow us to appreciate the variations in patient anxiety.
Change of Anxiety state(AE scale) | Before surgery and up to 2 hours after surgery
  The proportion of patients whose preoperative anxiety state (AE) is improved or stable between before and after the session with virtual reality headset. These two measurements will allow us to appreciate the variations in patient anxiety.

SECONDARY OUTCOMES:
Anxiety evaluation by Amsterdam Preoperative Anxiety and Information Scale (APAIS) | up to 1 month after surgery
  Anxiety score [minimum value 0 , up to maximum value (worse) 20] according to the Amsterdam Pre-operative Anxiety and Information Scale (APAIS)
Pain evaluation (Visual Analog Pain Scale) | up to 1 month after surgery
  Score on the VAS pain scale [minimum value 0, up to maximum value (worse) 10]
Satisfaction of patients by EVAN-G scale (Evaluation of the General Anesthesia feelings) | Up to 2 hours after surgery
  score of EVAN-G questionnaire [minimum value 0, up to maximum value (worse) 100]
Taking of anxiolytics | up to 1 month after surgery
  variation of amount of anti-anxiety medication

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre François Baclesse, Caen
  - CHU CAEN, Caen
  - Clinique Mathilde, Rouen

IPD SHARING:
Plan to Share IPD: No